CLINICAL TRIAL: NCT02986477
Title: Clinical Applications of Contrast-Enhanced Ultrasonography in Pediatric Population - Intravesicle Administration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00118038
Record Dates: First submitted 2016-12-05; First posted 2016-12-08 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Vesico-Ureteral Reflux
MeSH Terms: conditions — Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast Ultrasound (Other): Patients with vesicoureteral reflux will receive contrast ultrasound via Foley catheter for study of vesicoureteral reflux.
  Interventions: Other: Contrast Ultrasound

INTERVENTIONS:
Other: Contrast Ultrasound — For diagnostic purposes, intravesicle administration of contrast ultrasound agent will be performed to study vesicoureteral reflux.

SUMMARY:
In children, specifically the intravesicle administration to study vesicoureteral reflux in children already catheterized and scheduled for voiding cystourethrogram (VCUG). Contrast-enhanced ultrasonography is a tremendous advancement from conventional B-mode and color Doppler ultrasonography, as it permits noninvasive, non-ionizing delineation of physiology and pathophysiology with higher resolution and accuracy in children. The technique is particularly useful in pediatric population whose lifetime risk of cancer significantly increases with higher frequency of ionizing radiation. Voiding cystourethrogram is a fluoroscopy technique that can study reflux real time but at the risk of radiation side effects. In this regard, intravesicle administration of ultrasound contrast agent can help avoid radiation in children and potentially replace the conventionally used voiding cystourethrogram.

DETAILED DESCRIPTION:
The most commonly used genitourinary application of ultrasound contrast agent is for the diagnosis of vesicoureteral reflux via intra-vesicle administration of contrast agent. The utility of ultrasound contrast agent in contrast-enhanced voiding urosonography is well established and published over two decades (Darge 2002, Darge 2008, Darge 2010). As with other applications of ultrasound contrast agents, the method offers the advantages of no radiation, low cost, excellent anatomic detail, and higher sensitivity for reflux detection than VCUG. The most comprehensive study to detail the safety profile of intravesicle ultrasound contrast is by Papadopoulou et al. (Papadopoulou, Ntoulia et al. 2014) which described a total of 1,010 children (563 girls, 447 boys) with a mean age of 2.9 years. No adverse events were reported at 1 hour after exam. Follow-up phone interviews revealed no adverse events in the majority (973 of 1,010). The remaining 37 children experienced mild symptoms including dysuria (n=26) and urinary retention (n=2) which may have been related to catheterization rather than the contrast agent. A recent European survey at 29 centers evaluating the use of ultrasound contrast agent in 4,131 children for pediatric reflux diagnosis reported no adverse events (Riccabona 2012).

The procedure consists of pre-contrast, post-contrast, voiding phase, and post-void depiction of the kidneys, ureters, bladder, and transperineal scan of the urethra, for identification of potential ectopic ureters (Darge 2008, Duran, del Riego et al. 2012) that can easily be missed on non-distended ureters on CT, MRI, or radionuclide imaging. The two primary methods of contrast injection includes direct injection into a partially filled bladder (Darge 2008) and another using a saline bag for subsequent drip infusion via the catheter into the bladder (Back, Edgar et al. 2015).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 0-17 years undergoing an ultrasound for a clinical indication at the Johns Hopkins Hospital
* Willing to either extend a previously scheduled clinically indicated voiding cystourethrogram

Exclusion Criteria:

* Known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts
* History of hypersensitivity reactions to sulfur hexafluoride lipid microsphere components or to any of the inactive ingredients in LUMASON. Inactive ingredients include 1,2-Dipalmitoyl-sn-glycero-3-phosphoglycerol, sodium salt (DPPG), a minor (1-2%) component normally present in most cell membranes, Diasteroylphosphatidylcholine (DSPC), a commonly used synthetic phospholipids, and palmitic acid, the most commonly found fatty acid in animals.
* Patient subjects in unstable clinical condition.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Clinical Applications of Contrast-Enhanced Ultrasonography in Pediatric Population - Intravesicle Administration | 10 years
  The presence of vesicoureteral reflux is assessed as the primary outcome measure.
  Qualitative evaluation is performed to assess the presence of contrast within the collecting systems, which then correlates with vesicoureteral reflux.
  Since this is a qualitative evaluation based on the acquired radiologic images, there is no unit, but the degree of vesicoureteral reflux is assessed. Vesicoureteral reflux is graded into I to V grades based on the severity.

IPD SHARING:
Plan to Share IPD: No